CLINICAL TRIAL: NCT00322855
Title: Chart Review of Treatments Received by Patients Diagnosed With Soft Tissue Sarcoma
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0517C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chart Review: patients diagnosed with soft tissue sarcoma

SUMMARY:
To review the outcome of patients with soft tissue sarcoma treated with chemotherapy from 2004 and 2005.

DETAILED DESCRIPTION:
Chart review of patients with soft tissue sarcoma treated with chemotherapy from 2004 and 2005 to determine outcome

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with soft tissue sarcoma treated with chemotherapy form 2004 and 2005.

Exclusion Criteria:

* Not Specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with soft tissue sarcoma treated with chemotherapy form 2004 and 2005.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aroop Mangalik, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chart Review
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chart Review
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 17 [17 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: To Review the Outcome of Patients With Soft Tissue Sarcoma Treated With Chemotherapy From 2004 and 2005
Time Frame: up to one year
Population: Study was terminated due to low accrual. This is not an applicable trial; no results to report
Arm/Group | Chart Review
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed in this chart review study.
Arm/Group | Chart Review
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No